CLINICAL TRIAL: NCT07235592
Title: Post Market Clinical Follow-Up Study to Demonstrate the Safety and Performance of the PRESERFLO™ MicroShunt XI in Patients With Primary Open Angle Glaucoma
Brief Title: PRESERFLO™ MicroShunt XI Observational PMCF Study With no Control Group
Status: Not yet recruiting | Type: Observational
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: 200011001SW
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Primary Open Angle Glaucoma
Keywords: POAG
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Microshunt XI treatment group: MicroShunt XI will be surgically implanted in eyes of patients with primary open angle glaucoma where intra ocular pressure (IOP) remains uncontrollable while on maximum tolerated medical therapy and/or where glaucoma progression warrants surgery.
  Interventions: Device: Microshunt XI

INTERVENTIONS:
Device: Microshunt XI — The PRESERFLO™ MicroShunt XI is an implantable glaucoma drainage device
  Other Names: Intervention Model/Device: SIBS implant, OD 350 µm, lumen 71 µm, length 11 mm, triangular fins; subconjunctival/Tenon implantation.

SUMMARY:
The purpose of this study is to collect safety and performance data on the PRESERFLO™ MicroShunt XI in patients diagnosed with primary open angle glaucoma who are inadequately controlled on maximum tolerated medical therapy with intraocular pressure ≥18 mmHg and ≤35 mmHg and/or where glaucoma progression warrants surgery.

DETAILED DESCRIPTION:
This is a prospective, multicentric, single arm post market clinical follow-up study to collect safety and performance data on the CE Marked PRESERFLO™ MicroShunt XI device in patients with primary open angle glaucoma. The PRESERFLO™MicroShunt XI employs a tube to create a conduit for the flow of aqueous humor from the anterior chamber of the eye to a bleb formed under the conjunctiva and Tenon's capsule; the front/ proximal end of the tube extends into the anterior chamber while the back/ distal end terminates in the bleb. The PRESERFLO™MicroShunt XI reduces IOP by physically shunting aqueous humor from the high pressure anterior chamber to the lower pressure bleb. The intended users of the PRESERFLO™ MicroShunt XI are ophthalmologists/ophthalmic surgeons specialized in the treatment of glaucoma (including surgeons specialized in anterior segment and cataract surgery) who have been trained to use the device. No biospecimens are collected in this study and no control group.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 85 years, inclusive
2. Patient diagnosed with primary open glaucoma where the IOP is not adequately controlled on maximum tolerated medical therapy and has intraocular pressure ≥18 mmHg and ≤35 mmHg while on glaucoma medications
3. Patient willing to comply with study requirements
4. Patient who has signed an approved informed consent form

Exclusion Criteria:

1. Angle closure glaucoma
2. Presence of conjunctival scarring, previous incisional ophthalmic surgery involving the conjunctiva or conjunctival pathologies (e.g., thin conjunctiva, pterygium)
3. Active iris neovascularization
4. Active inflammation (e.g., blepharitis, conjunctivitis, scleritis, keratitis, uveitis)
5. Vitreous in the anterior chamber
6. Presence of an anterior chamber intraocular lens (ACIOL)
7. Intraocular silicone oil
8. Need for glaucoma surgery combined with other ocular procedures (e.g., cataract surgery with IOL implantation) or anticipated need for additional ocular surgery during the investigational period
9. Central corneal thickness that is less than 450 microns or greater than 620 microns
10. Previous cilioablative procedure
11. Neovascular glaucoma
12. Uveitic Glaucoma
13. Pseudoexfoliative or pigmentary glaucoma
14. Chronic inflammation
15. Previous incisional ophthalmic surgery within 6 months prior to study
16. Enrolled in this or another study (only one eye can participate in this study) or completed their participation in another study within 30 calendar days of the screening exam
17. Ocular pathology or medical condition for which, in the investigator's judgment, the following factors would either place the patient at increased risk of complications or contraindicate device implantation or interfere with compliance to elements of the Protocol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients with primary open angle glaucoma where IOP remains uncontrollable while on maximum tolerated medical therapy and/or where glaucoma progression warrants surgery. At the time of a scheduled clinic visit, eligible patients will be invited to participate in the study and willing patients will be requested to sign an informed consent form. Once informed consent is obtained, the subject is included in the study and relevant data will be recorded during scheduled clinical visits. Participation in this study is entirely voluntary;
Sampling Method: Non-Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Primary Performance Outcome to determine the change in the proportion of eyes with change in intraocular pressure | Screening to 12 months
  This is a primary performance outcome to determine the proportion of eyes with ≥20% change and 6 mmHg to <21 mmHg intraocular pressure from screening to 12 months

SECONDARY OUTCOMES:
Secondary Performance Outcome to determine the change in the proportion of eyes with change in intraocular pressure | At 12 months
  This is a secondary performance outcome to determine the proportion of eyes with ≥20% change and 6 mmHg to <18 mmHg intraocular pressure at 12 months

OTHER OUTCOMES:
Primary Safety Outcome Incidence of all device- and/or procedure-related adverse events | Screening to 12 months
  This is a primary safety outcome for Incidence of all device- and/or procedure-related adverse events during the study

CONTACTS AND LOCATIONS:
Locations (11):
- AKH Wien, Vienna, Austria
- Glaucoma Clinic, UZ Leuven, Leuven, Belgium
- Germany (2):
  - Internationale Innovative Opthalmochirurgie GbR, Düsseldorf
  - Universitätsklinikum Tübingen, Department für Augenheilkunde, Tübingen
- Italy (2):
  - Irccs Fondazione G. B. Bietti, Rome
  - Policlinico Universitario Molinette, Turin
- Universiteitskliniek voor Oogheelkunde Maastricht, Maastricht, Netherlands
- ULS Santa Maria, Lisboa, Lisbon, Portugal
- Hospital Clinico San Carlos, San Carlos, Spain
- United Kingdom (2):
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - Moorfields Eye Hospital NHS Foundation Trust, London